CLINICAL TRIAL: NCT03740893
Title: PHOENIX DDR/Anti-PD-L1 Trial: A Pre-surgical Window of Opportunity and Post-surgical Adjuvant Biomarker Study of DNA Damage Response Inhibition With or Without Anti-PD-L1 Immunotherapy in Patients With Neoadjuvant Treatment Resistant Residual Triple Negative Breast Cancer
Acronym: PHOENIX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICR-CTSU/2017/10065; 2018-002077-21 (EudraCT Number); ISRCTN47127434 (Registry Identifier: ISRCTN Registry); CRUKE/16/026 (Other: Cancer Research UK)
Record Dates: First submitted 2018-10-05; First posted 2018-11-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasm; Triple Negative Breast Cancer (TNBC); HRD
Keywords: AZD6738; Olaparib; Durvalumab; Window of opportunity; Triple negative breast cancer; Breast cancer; Homologous Repair Deficiency (HRD)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — ceralasertib; olaparib; durvalumab

STUDY DESIGN:
Intervention Model Description: WOP, open-label, multi-centre, phase IIa trial comprising multiple non-comparative treatment cohorts with patient allocation via minimisation (cohorts A-D) or allocation according to HRD and germline BRCA1/2 mutation status (cohorts E-G).
  The trial consists of two parts: a post-neoadjuvant treatment preoperative WOP component (PART 1); and a post-operative component (PART 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort A (standard care reference cohort) (No Intervention): Arm formally closed to recruitment since 06 August 2024
- Cohort B (AZD6738 monotherapy) (Experimental): Arm formally closed to recruitment since 06 August 2024
  Interventions: Drug: AZD6738
- Cohort C (olaparib monotherapy) (Experimental): Arm formally closed to recruitment since 06 August 2024
  Interventions: Drug: Olaparib
- Cohort D (durvalumab monotherapy) (Experimental): Arm formally closed to recruitment since 06 August 2024
  Interventions: Drug: Durvalumab
- Cohort E: non-HRD and gBRCA1gBRCA1/2 wildtype confirmed at HRD screening (Experimental)
  Interventions: Drug: Olaparib
- Cohort F: gBRCA1/2 mutation confirmed at HRD screening (Experimental)
  Interventions: Drug: Olaparib; Drug: Durvalumab
- Cohort G: HRD & gBRCA1/2 wildtype confirmed at HRD screening (Experimental)
  Interventions: Drug: Olaparib; Drug: Durvalumab

INTERVENTIONS:
Drug: AZD6738 — PART 1: Pre-operative exposure of 160mg AZD6738 to be administered orally twice daily on Days 5 -14 of the WOP.
  PART 2: 12 months post-operative exposure to 160mg AZD6738 to be administered orally twice daily on Days 1 - 14 of a 28 day cycle.
  AZD6738 was removed as intervention under investigation as of 06 August 2024 (due to formal closure of cohort B)
  Arms: Cohort B (AZD6738 monotherapy)
Drug: Olaparib — PART 1 (cohort C, and cohorts E-G): Pre-operative exposure to 300mg of olaparib to be administered orally twice daily on Days 1-14 of the WOP.
  PART 2 (cohort C, and cohorts F and G): 12 months post-operative exposure to 300mg olaparib (2 x 150mg tablets) to be administered orally twice daily on a continuous schedule Day 1-28 of a 28 day cycle.
  Cohort C was formally closed to recruitment since 06 August 2024.
  Arms: Cohort C (olaparib monotherapy); Cohort E: non-HRD and gBRCA1gBRCA1/2 wildtype confirmed at HRD screening; Cohort F: gBRCA1/2 mutation confirmed at HRD screening; Cohort G: HRD & gBRCA1/2 wildtype confirmed at HRD screening
Drug: Durvalumab — PART 1 (cohort D): Pre-operative exposure to 1500mg durvalumab to be administered via intravenous (IV) infusion on Day 1 only of the WOP.
  PART 2 (cohorts A and D, and cohorts F and G): 12 months post-operative exposure to 1500mg durvalumab to be administered via intravenous (IV) infusion on Day 1 only of a 28 day cycle.
  Cohorts A and D were formally closed to recruitment since 06 August 2024.
  Arms: Cohort D (durvalumab monotherapy); Cohort F: gBRCA1/2 mutation confirmed at HRD screening; Cohort G: HRD & gBRCA1/2 wildtype confirmed at HRD screening

SUMMARY:
PHOENIX is a window of opportunity (WOP), open-label, multi-centre, phase IIa trial comprising multiple non-comparative treatment cohorts with patient allocation via minimisation (cohorts A-D) or allocation according to HRD and germline BRCA1/2 mutation status (cohorts E-G). The trial consists of two parts: a post-neoadjuvant treatment preoperative WOP component (PART 1); and a post-operative component (PART 2).

Cohorts A-D: To assess whether short exposure to a DDR inhibitor or anti-PD-L1 immunotherapy in a preoperative WOP in patients with post-NACT high risk residual disease, generates a signal of anti-tumour biological activity within residual disease tissue.

Cohort E: To assess whether short exposure to a DDR inhibitor with or without anti-PD-1 immunotherapy in a preoperative WOP in patients with non-HRD associated TNBC and post-neoadjuvant treatment high risk residual disease, generates a signal of anti-tumour biological activity within residual disease tissue.

Cohorts F & G: To assess whether short exposure to the DDR inhibitor olaparib with or without anti-PD-1 immunotherapy in a preoperative WOP in patients with HRD associated TNBC and post-neoadjuvant treatment high risk residual disease, generates a signal of anti-tumour biological activity within residual disease tissue.

DETAILED DESCRIPTION:
Cohorts A-D have been formally closed for recruitment since 06 August 2024.

ELIGIBILITY:
Inclusion Criteria for Trial Registration:

1. Signed Informed Consent Form (ICF) for Trial Registration;
2. Aged ≥18 years old;
3. Histologically confirmed invasive triple negative breast cancer (TNBC). TNBC defined as ER negative, PgR negative (ER and PgR negative as defined by Allred score 0/8, 1/8 or 2/8 or stain in <1% of cancer cells) or PgR unavailable, and HER2 negative (immunohistochemistry 0/1+ or negative in situ hybridization) as determined by local laboratory and recorded in the patients notes;
4. Planned definitive surgical treatment after at least 6 cycles of neoadjuvant chemotherapy (NACT) Patients currently receiving SOC pembrolizumab, or having previously received SOC pembrolizumab but subsequently discontinued treatment, in combination with NACT are eligible for Trial Registration;
5. Radiographically measurable tumour mass assessable for new distinct radio-opaque marker insertion and repeated biopsies on the NACT mid-assessment standard of care imaging modality;
6. Eastern Oncology Cooperative Group (ECOG) performance status 0-1;
7. Considered fit enough to have breast cancer surgery with curative intent;
8. Considered fit to complete at least 2 weeks of pre-operative trial treatment in the WOP;
9. Patients must be suitable for a mandatory pre-treatment baseline biopsy performed Day -1 or 1 of the window of opportunity (WOP) and a post-treatment biopsy performed on Day 14 of the WOP. Registered patients who are approached for Trial Entry will be required to consent to the pre- and post- WOP treatment biopsy. If it is deemed unsafe to proceed with biopsy upon Trial Entry the patient will not be eligible for participation in the trial.
10. Patients with clinical stage II or III disease or clinical suspicion of metastatic disease must have staging studies to exclude metastatic disease if this is standard of care, and staging methods should be used as per standard of care (axillary lymph nodes or internal mammary node involvement will not be regarded as evidence of metastatic disease);
11. Patients with previous invasive cancers (including breast cancer) are eligible if the treatment was completed >5 years prior to Trial Registration, and there is no evidence of recurrent disease;
12. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up schedule; those conditions should be discussed with the patient before Trial Registration;
13. Patients must be a) surgically sterile (i.e. if female have undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy; if male have undergone a bilateral orchidectomy); b) have a sterilised sole partner; or c) be post-menopausal; or d) must agree to practice total/true abstinence; or e) use a condom and one highly effective form of contraception in combination during the period of trial treatment and be willing to do so for a period of at least 6 months following the end of trial treatment. Please refer to Section 5.4 Lifestyle Guidance for the definition of total/true abstinence and a list of the permitted highly effective forms of contraception.

Post-menopausal is defined by at least one of the following criteria:

1. Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
2. Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution for women < 50 years of age not using hormonal contraception or hormonal replacement therapy. Please note: in absence of amenorrhea for 1 year, a single LH and/or FSH measurement is insufficient.
3. Radiation-induced oophorectomy with last menses >1 year ago
4. Chemotherapy-induced menopause with >1 year interval since last menses
5. Surgical sterilisation (hysterectomy, bilateral salpingectomy or bilateral oophorectomy)

Exclusion Criteria for Trial Registration:

1. Definitive evidence of metastatic disease (axillary lymph nodes or internal mammary node involvement will not be regarded as evidence of metastatic disease) ;
2. Patients with bilateral tumours.
3. History of another primary malignancy within the last 5 years prior to Trial Registration, except for:

   1. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease;
   2. Adequately treated carcinoma in situ without evidence of disease;
4. Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML;
5. Severe concurrent disease, infection or co-morbidity that, in the judgment of the local Investigator, would make the patient inappropriate for Trial Registration;
6. Resting ECG indicating uncontrolled, potentially irreversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >470 msec, electrolyte disturbances, etc.), or patients with congenital long QT syndrome;
7. Patients unable to swallow orally administered medication;
8. Patients receiving therapeutic anti-coagulation treatment (including warfarin and novel oral anti-coagulants).
9. Patients with gastrointestinal disorder affecting absorption (e.g. gastrectomy, active peptic ulcer disease within last 3 months);
10. History of seizure or any condition that may predispose to seizure.
11. Other non-malignant systemic disease that would preclude trial treatment or would prevent required follow-up;
12. Pregnant or breast-feeding;
13. Prior exposure to PARP inhibitor, including olaparib, anti-PD-1 or anti-PDL1 immunotherapy (including durvalumab) except for pembrolizumab if received as standard of care in combination with neoadjuvant chemotherapy;
14. Any other disease(s), psychiatric condition, metabolic dysfunction, or findings from a physical examination or clinical laboratory test result that in the investigators opinion would cause reasonable suspicion of a disease or condition, that contraindicates the use of trial treatment, that may increase the risk associated with trial participation, that may affect the interpretation of the results, or that would make this trial inappropriate for the patient;
15. Patients with a known hypersensitivity to pembrolizumab, durvalumab or olaparib or any excipients of the products;
16. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT);
17. Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (HBV; known positive HBV surface antigen (HBsAg) result), hepatitis C (HCV), or human immunodeficiency virus (HIV; positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA;

Inclusion Criteria for Trial Entry:

1. Signed Informed Consent Form (ICF) for Trial Entry;
2. Residual disease is confirmed as at least one viable disease focus ≥1cm on trial-specific imaging performed at least 1 week following day 1 of the final cycle of NACT.
3. Provision of acceptable archival diagnostic tumour tissue sample prior to Trial Entry as defined in the Investigator Laboratory Manual.
4. Recovery from all acute adverse events of prior NACT or pembrolizumab to baseline or NCI CTCAE Grade ≤1, except for alopecia. Patients with irreversible toxicity not reasonably expected to be exacerbated by trial treatment may be included only after consultation with the CI or Coordinating Investigator.
5. Patients must have adequate haematological, renal and hepatic function as defined by:

   * Haemoglobin (Hb) ≥ 10 g/dL (≥ 100 g/L) with no blood transfusion in the past 28 days
   * Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 x 109/L)
   * Platelet count ≥100,000/mm3 (≥ 100 x 109/L)
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional ULN
   * Calculated creatinine clearance ≥51 mL/min using the Cockcroft-Gault equation (please refer to Appendix 4) or based on a 24 hour urine test or another validated test as per local practice
6. Women of childbearing potential must have a confirmed menstrual period and a negative urinary or serum pregnancy test prior to Trial Entry. This should be repeated as applicable to ensure a negative pregnancy test is performed on the day of planned trial treatment.
7. Confirmation that all Trial Registration inclusion criteria listed in Section 5.3.1 remain satisfied.

Exclusion Criteria for Trial Entry:

1. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
2. Major surgery (excluding minor procedures, e.g. placement of vascular access) within 2 weeks prior to Trial Entry. Patients must have recovered from any effects of any major surgery prior to commencing trial treatment.
3. Use of any investigational agent within 30 days prior to commencing trial treatment.
4. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to commencing trial treatment is 5 weeks;
5. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (e.g. bosentan, efavirenz, modafinil) CYP3A inducers. The required washout period prior to commencing trial treatment is 5 weeks;
6. Whole blood infusion within 28 days prior to trial entry (packed red blood cells and platelet transfusions are acceptable).
7. Receipt of live attenuated vaccine within 30 days prior to commencing trial treatment.
8. Confirmation that none of the Trial Registration exclusion criteria listed in Section 5.3.2 are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Cohorts B and C co-primary endpoint #1: Change in mean proliferation index (as measured by tumour cell Ki67 staining) post WOP intervention within post-treatment biopsy compared to pre-treatment baseline biopsy. | Post 2 weeks of trial treatment in the window of opportunity
  Change in mean proliferation index (as measured by tumour cell Ki67 staining) post WOP intervention within post-treatment biopsy compared to pre-treatment baseline biopsy. A patient will be defined as being a Ki67 responder if they experience a relative decrease in Ki67 positive cells of ≥33% in the post-treatment biopsy sample. This represents a characterised threshold that we do not believe would be exceeded by chance in this patient population.
  AND/OR Cohorts B and C co-primary endpoint #2, as described below.
Cohorts B and C co-primary endpoint #2: Changes in the proliferation gene expression signature post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy. | Post 2 weeks of trial treatment in the window of opportunity
  Changes in the proliferation gene expression signature post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy. A patient will be defined as being a responder if there is a ≥1.5-fold drop in the proliferation gene expression in the surgical resection sample.
  The proliferation gene signature will be based on this list of 11 highly correlated proliferation genes shown in multiple studies including those published by The Cancer Genome Atlas and they also contribute to the calculation of the proliferation score in the publicly available PAM50 classifier. The list consists of :"CCNB1","UBE2C","BIRC5","NDC80","CDC20","PTTG1","RRM2","MKI67","TYMS","CEP55","NUF2"
  For each sample, a proliferation gene module score will be calculated according to the expression of the relevant genes.
  AND/OR Cohorts B and C co-primary endpoint #1, as described above.
Cohort D co-primary endpoint #1: Change in frequency of CD8+ sTILs post anti-PD-L1 immunotherapy within the post-treatment biopsy compared to pre-treatment baseline biopsy. | Post 2 weeks of trial treatment in the window of opportunity
  Change in frequency of CD8+ sTILs post anti-PD-L1 immunotherapy within the post-treatment biopsy compared to pre-treatment baseline biopsy. A patient will be defined as being a responder if they experience an absolute increase of ≥ 10% in the percentage CD8+ sTILs within the post-treatment biopsy sample.
  The % CD8+ sTILs value denotes the area occupied by CD8+ sTILs over total intratumoural stromal area.
  AND/OR Cohort D co-primary endpoint #2, as described below.
Cohort D co-primary endpoint #2: Changes in the interferon gamma-positive (IFNγ+) signature post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy. | Post 2 weeks of trial treatment in the window of opportunity
  Changes in the interferon gamma-positive (IFNγ+) signature post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy. A patient will be defined as being a responder if there is a ≥2-fold increase in the IFNγ+ gene expression in the post-treatment biopsy sample.The four-gene IFNγ+ score will be calculated, comprising of IFNγ, CD274, LAG3, and CXCL9.
  AND/OR Cohort D co-primary endpoint #1, as described above.
Cohorts F and G co-primary endpoint #1: Change in mean proliferation index (as measured by tumour cell Ki67 staining) post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy. | Post 2 weeks of trial treatment in the window of opportunity
  Change in mean proliferation index (as measured by tumour cell Ki67 staining) post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy.
  A patient will be defined as being a Ki67 responder if they experience a relative decrease in Ki67 positive cells of ≥33% in the post-treatment biopsy sample. This represents a characterised threshold that we do not believe would be exceeded by chance in this patient population.
  AND/OR Cohorts F and G co-primary endpoints #2 and #3, as described below
Cohorts F and G co-primary endpoint #2: Changes in the proliferation gene expression signature post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy. | Post 2 weeks of trial treatment in the window of opportunity
  Changes in the proliferation gene expression signature post WOP intervention within the post-treatment biopsy compared to pre-treatment baseline biopsy.
  A patient will be defined as being a responder if there is a ≥1.5-fold drop in the proliferation gene expression in the post-treatment biopsy sample.
  The proliferation gene signature will be based on this list of 11 highly correlated proliferation genes shown in multiple studies including those published by The Cancer Genome Atlas and they also contribute to the calculation of the proliferation score in the publicly available PAM50 classifier. The list consists of : "CCNB1","UBE2C","BIRC5","NDC80","CDC20","PTTG1","RRM2","MKI67","TYMS","CEP55","NUF2"
  For each sample, a proliferation gene module score will be calculated according to the expression of the relevant genes.
  AND/OR Cohorts F and G co-primary endpoints #1 and #3, as described above, and below respectively
Cohorts F and G co-primary endpoint #3: Changes in the plasma ctDNA (D0-D14) post WOP intervention compared to pre-treatment. | Post 2 weeks of trial treatment in the window of opportunity
  Changes in the plasma ctDNA (D0-D14) post WOP intervention compared to pre-treatment.
  A patient will be defined as being a responder if the ratio of ctDNA post-WOP compared to pre-WOP is <0.25. This cut-off has been selected in line with other studies of PARP inhibitors in TNBC.
  AND/OR Cohorts F and G co-primary endpoints #1 and #2, as described above

SECONDARY OUTCOMES:
Incidence of adverse events during trial treatment | 1 month post-surgery
  Incidence of adverse events (AEs) during trial treatment (including surgical complications) by treatment cohort at 1 month post-surgery.
Response in cohort E | Post 2 weeks of trial treatment in the window of opportunity
  Response in Cohort E, defined as per the co-primary endpoints for cohorts F-G.
Methylation status of BRCA1 and RAD51C | Post 2 weeks of trial treatment in the window of opportunity
  Methylation status (methylated vs. non-methylated and level of methylation) of BRCA1 and RAD51C on diagnostic and pre- and post-WOP tumour samples and changes in methylation levels between these timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tutt, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (6):
- United Kingdom (6):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - King's College Hospital, London, England
  - Christie Hospital NHS Trust, Manchester, England
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - Guy's and St Thomas' Hospital NHS Foundation Trust, London
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No